CLINICAL TRIAL: NCT00528151
Title: A Randomized, Double-blind, Placebo-controlled Trial of Curcumin in Leber's Hereditary Optic Neuropathy (LHON)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123/2547
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2004-08

CONDITIONS: Optic Atrophy, Hereditary, Leber
Keywords: Curcumin, LHON, antioxidant, visual outcome
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Placebo Comparator): 1. curcumin
  2. placebo
  Interventions: Drug: curcumin

INTERVENTIONS:
Drug: curcumin — curcumin 250 mg twice a day in the first group. placebo 1 capsule twice a day in the second group.

SUMMARY:
Background Leber's Hereditary Optic Neuropathy (LHON) is a maternally inherited ocular disorder associated with a mutation in mtDNA . The common manifestation is visual loss which caused by the respiratory chain enzymes complex dysfunction resulting in increased oxidative stress enzymes production.

Purpose To determine whether curcumin which is an antioxidant agent is beneficial to the patients with 11778 LHON mutation.

Material and Method Seventy patients with 11778 LHON mutation were randomly treated with oral curcumin (500 mg/day) and placebo for 1 year. The visual acuity, computerized visual field, electrophysiologic parameters and oxidative stress enzymes in plasma were compared before and after treatment at 3, 6, and 12 months interval.

DETAILED DESCRIPTION:
Leber's hereditary optic neuropathy (LHON) is a maternally inherited disease that is characterized by a simultaneous or more common sequential bilateral loss of central vision, which typically occurs during the teenager years or early adulthood. The disease may be progressive and the patients eventually become blind. In contrast to blindness in patients caused by congenital diseases, the patients who develop blindness caused by LHON will have more trouble in their life because they previously had better vision. Although LHON is associated with mitochondrial DNA mutation at a variable nucleotide position but no certain mechanism of optic nerve injury has been found. It has been postulated that a defect in a complex of respiratory chain enzyme which is caused by mitochondrial DNA dysfunction, results in an increase of free radical substances that interfere with optic nerve function in LHON. Some antioxidant substances have been used to decrease the progression of visual impairment. However, there have been few therapeutic trials for LHON.

Curcumin, a component of tumeric, which comes from the root Curcumin longa has antioxidant, anti-inflammatory and anti-carcinogenic activities. There is some evidence which suggests that curcumin contributes to the in vitro removal of free radical gradients in thalassemic serum and to a clinical improvement of thalassemic patients. We propose a randomized controlled trial study of curcumin, which is an antioxidant substance, for LHON. This study will provide not only an insight into the therapeutic efficacy of curcumin, a kind of Thai herb, for LHON but also the development of future therapeutic strategies to prevent blindness.

ELIGIBILITY:
Inclusion Criteria:

* LHON patient with 11778 point mutation

Exclusion Criteria:

* LHON patient with other point mutation

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-05; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
visual outcome | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Professor Wanicha L Chuenkongkaew, MD, Principal Investigator — Mahidol University
Locations (1):
- Professor Wanicha Chuenkongkaew, Bangkok, Bangkok, Thailand